CLINICAL TRIAL: NCT02411773
Title: Functional Sympatholysis and Exercise Intolerance in Chronic Kidney Disease
Brief Title: Sympatholysis in Chronic Kidney Disease
Acronym: Sym-CKD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jeanie Park, Associate Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00078214
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium Bicarbonate; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Exercise Training plus Sodium Bicarbonate (Active Comparator): Subjects with CKD will undergo exercise training on a stationary bicycle for 20-45 minutes, 3 times per week, for 6-12 weeks. Additionally, subjects will take 1300-2600 mg (2-4 pills) of sodium bicarbonate prior to each exercise session three times a week.
  Interventions: Drug: Sodium Bicarbonate; Behavioral: Exercise Training
- Exercise Training plus Placebo (Active Comparator): Subjects with CKD will undergo exercise training on a stationary bicycle,for 20-45 minutes, 3 times per week, for 6-12 weeks. Additionally, subjects will take 2-4 placebo tablets prior to each exercise session three times a week.
  Interventions: Drug: Placebo; Behavioral: Exercise Training
- Control to Exercise (Stretching) plus Sodium Bicarbonate (Active Comparator): Subjects with CKD will undergo progressive whole body stretching and toning exercises 3 times a week for 20-45 minutes for 6-12 weeks. Additionally, subjects will take 1300-2600 mg (2-4 pills) of sodium bicarbonate prior to each stretching session three times a week.
  Interventions: Drug: Sodium Bicarbonate; Behavioral: Control to Exercise (Stretching)
- Control to Exercise (Stretching) plus Placebo (Placebo Comparator): Subjects with CKD will undergo progressive whole body stretching and toning exercises 3 times a week for 20-45 minutes for 6-12 weeks. Additionally, subjects will take 2-4 placebo tablets prior to each exercise session three times a week.
  Interventions: Drug: Placebo; Behavioral: Control to Exercise (Stretching)
- Healthy Control (No Intervention): Healthy subjects without CKD will not receive any interventions.

INTERVENTIONS:
Drug: Sodium Bicarbonate — Sodium bicarbonate tablet is 650 mg for one tablet. Oral sodium bicarbonate will be given out as 1300mg-2600mg (2-4 pills) prior to each exercise or stretching session. Serum bicarbonate measurements will be monitored throughout the study (at 2 weeks, then every 2-4 weeks thereafter), and bicarbonate dosages will be adjusted to avoid metabolic alkalosis (serum bicarbonate > 30).
  Arms: Control to Exercise (Stretching) plus Sodium Bicarbonate; Exercise Training plus Sodium Bicarbonate
Drug: Placebo — 2-4 placebo pills will be given out prior to each exercise or stretching session.
  Arms: Control to Exercise (Stretching) plus Placebo; Exercise Training plus Placebo
Behavioral: Exercise Training — Exercise training consists of riding a stationary bicycle for 20-45 minutes, 3 times per week, supervised by trained exercise specialists, for 6-12 weeks. The exercise program will follow the guidelines provided by the American College of Sports Medicine (ACSM) for optimizing cardiovascular fitness. Exercise intensity will begin at low levels (50 percent of resting heart rate) and increase to no greater than 80 percent of resting heart rate. Exercise time will progress, depending on subject's progress, from 20 minutes per session at first, to a maximum of 45 minutes. Trained staff members will give instructions throughout each exercise session. Before beginning each exercise session, subjects will be instructed on a warm-up focusing on preparing the legs for activity.
  Arms: Exercise Training plus Placebo; Exercise Training plus Sodium Bicarbonate
Behavioral: Control to Exercise (Stretching) — Stretching exercise will consist of muscle stretching and toning for 20-45 minutes, 3 times per week, supervised by trained exercise specialists, for 6-12 weeks. Trained staff members will guide subjects with the stretching exercises, and activities are designed to increase flexibility and range of motion. Before beginning each stretching exercise session, subjects will be instructed to warm-up.
  Arms: Control to Exercise (Stretching) plus Placebo; Control to Exercise (Stretching) plus Sodium Bicarbonate

SUMMARY:
The purpose of this study is to find out why patients with chronic kidney disease (CKD) have poor exercise capacity and what causes an increase in blood pressure during exercise (i.e. increased adrenaline levels, or decreased ability of blood vessels to dilate).

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) suffer from exercise intolerance and poor physical capacity which contributes to increased cardiovascular risk in this patient population. Prior studies have shown that CKD patients have an exaggerated increase in blood pressure (BP) during both static and rhythmic exercise. Such abnormal hemodynamic responses to exercise can contribute to poor physical capacity and abnormal muscle blood flow during exercise in these patients. The goals of this project are to investigate the mechanisms and potential therapies targeting the abnormal hemodynamic response during exercise in CKD by examining the roles of impaired vasodilation, and exaggerated vasoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with Stages III and IV Chronic Kidney Disease (CKD)
* Kidney transplant recipients with varying degrees of kidney function
* Veterans 18-75 years old, without kidney disease, as study controls
* Exercise less than 20 minutes twice per week
* Willing and able to cooperate with the protocol

Exclusion Criteria:

* Severe CKD (estimated glomerular filtration rate (eGFR) < 15 cc/minute)
* Metabolic alkalosis (serum bicarbonate > 28 meq/L)
* Ongoing drug or alcohol abuse
* Diabetic neuropathy
* Any serious systemic disease that might influence survival
* Severe anemia with hemoglobin (Hbg) level < 10 g/dL
* Clinical evidence of congestive heart failure or ejection fraction below 35%
* Symptomatic heart disease determined by prior electrocardiogram, stress test, and/or history
* Treatment with central alpha agonists (clonidine)
* Uncontrolled hypertension with blood pressure (BP) greater than 170/100 mmHg
* Low blood pressure with BP less than 100/50 mmHg
* Pregnancy or plans to become pregnant
* Current treatment with monoamine oxidase inhibitors (MAOIs)
* Inability to exercise on a stationary bicycle

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-06-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in muscle oxygenation after exercise/stretching training | Baseline, Week 12
  Near-infrared spectroscopy (NIRS) will measure and record tissue oxyhemoglobin, deoxyhemoglobin, and total hemoglobin.
Change in muscle interstitial pH after exercise/stretching training | Baseline, Week 12
  Near-infrared spectroscopy (NIRS) will give an estimation of the pH levels within the muscle interstitial space. Muscle interstitial pH markedly decreases during exercise, and is often lower than blood pH with a larger intracellular to interstitial pH gradient. CKD patients may have less ability to buffer pH changes in the interstitial space during exercise. Bicarbonate supplementation may improve muscle interstitial buffering capacity during exercise, and prevent exaggerated reductions in muscle interstitial pH during exercise.
Change in venoconstriction after exercise/stretching training | Baseline, Week 12
  Dorsal hand vein model will be used to assess vascular alpha-1 adrenergic responsiveness by measuring the degree of venous constriction in response to varying dosages of local phenylephrine (PE) infusion.

SECONDARY OUTCOMES:
Change in Functional Sympatholysis | Baseline, 30 minutes
  Functional sympatholysis is determined by measuring the change in forearm oxygenation via near infrared spectroscopy (NIRS), and forearm blood flow and conductance using ultrasound, during sympathetic activation induced by lower body negative pressure (LBNP), at rest and during handgrip exercise. NIRS measures and records tissue oxyhemoglobin, deoxyhemoglobin, and total hemoglobin.
Change in muscle interstitial pH after handgrip exercise | Baseline, 30 minutes
  Near-infrared spectroscopy (NIRS) will give an estimation of the pH levels within the muscle interstitial space. Muscle interstitial pH markedly decreases during exercise, and is often lower than blood pH with a larger intracellular to interstitial pH gradient. CKD patients may have less ability to buffer pH changes in the interstitial space during exercise. Bicarbonate supplementation may improve muscle interstitial buffering capacity during exercise, and prevent exaggerated reductions in muscle interstitial pH during exercise.
Change in Venoconstriction after Phenylephrine | Baseline, 30 minutes
  Vascular function is measured as venoconstriction after administration of phenylephrine. Dorsal hand vein model will be used to assess vascular alpha-1 adrenergic responsiveness by measuring the degree of venous constriction in response to varying dosages of local phenylephrine (PE) infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanie Park, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No